CLINICAL TRIAL: NCT04269642
Title: Phase IIa Study to Evaluate the Efficacy and Safety of Subcutaneous SR-Exenatide (PT320) in Patients With Early Parkinson's Disease
Brief Title: SR-Exenatide (PT320) to Eveluate Efficacy and Safety in Patients With Early Parkinson's Disease
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Peptron, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PT320-201
Record Dates: First submitted 2020-01-13; First posted 2020-02-17 (Actual); Last update posted 2021-04-12 (Actual); Status verified 2021-04

CONDITIONS: Early Parkinson's Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- PT320 2.0mg Placebo (Placebo Comparator): will be injected subcutaneously once a week for 48 weeks
  Interventions: Drug: PT320 2.0mg Placebo
- PT320 2.0mg treatment 1 (Experimental): will be injected subcutaneously once a week for 48 weeks
  Interventions: Drug: PT320 2.0 mg
- PT320 2.5mg treatment2 (Experimental): will be injected subcutaneously every two weeks for 48 weeks. (Actually, patients will be injected PT320 2.5 mg and placebo alternately once a week.)
  Interventions: Drug: PT320 2.5 mg

INTERVENTIONS:
Drug: PT320 2.0mg Placebo — PT320 2.0mg Placebo
  Arms: PT320 2.0mg Placebo
Drug: PT320 2.0 mg — Exenatide slowly released formulation
  Arms: PT320 2.0mg treatment 1
Drug: PT320 2.5 mg — Exenatide slowly released formulation
  Arms: PT320 2.5mg treatment2

SUMMARY:
This study is to evaluate the safety and efficacy of sustained release (SR)-Exenatide (PT320, Q1W and Q2W) in the treatment of patients with early Parkinson's disease (PD).

DETAILED DESCRIPTION:
This study is a multicenter, randomized, double-blind, placebo-controlled, parallel comparison, phase IIa clinical study to evaluate the efficacy and safety of sustained release (SR)-Exenatide (PT320) in the treatment of patients with early Parkinson's disease (PD).

Exenatide (GLP-1) has been approved by the Food and Drug Administration (FDA) to treat patients with Type 2 Diabetes (T2D) and obesity. In addition, several research groups have confirmed that Exenatide has beneficial aspects due to the neuroprotective effects in neuronal cells in patients with PD. Peptron has developed a sustained-release (SR)-Exenatide, (PT320, Q1W and Q2W), which has shown a higher Blood-Brain Barrier (BBB) penetration rate and better patient compliance.

Thus, the objective of this study is to evaluate the effect of PT320 on symptom improvement and the inhibition of disease progression in the treatment of patients with early Parkinson's disease. Also, pharmacokinetic analysis of PT320 in blood cerebrospinal fluid (CSF) and exosome analysis of biomarkers related to Exenatide will be being tested, as exploratory measurements.

ELIGIBILITY:
Inclusion Criteria:

1. Patient who is male or female aged 40-75 and is diagnosed with Parkinson's Disease (using Queen Square Brain Bank criteria)
2. Patient who is diagnosed of Parkinson's Disease less than 24 months prior to the screening
3. Patient who has a modified Hoehn and Yahr stage ≤ 2. 5
4. Patient who has been taking L-dopa stable-dose less than 600 mg/day or who has not previously taken any medication for the treatment of Parkinson's Disease from 4 weeks prior to the screening.
5. Patient who is able to inject an Investigational Product by himself/herself or a his/her guardian.
6. Patient or legally acceptable representative who signs the informed consent form voluntarily and is able to comply with all study procedures

Exclusion Criteria:

1. Patient who is diagnosed or suspected to have Parkinson-plus syndromes (e.g., Multiple System Atrophy, Progressive Supranuclear Palsy, Corticobasal Degeneration, Diffuse Lewy Body Disease, and etc.)
2. Patient who has a BMI < 18.5 at the screening
3. Patient who has known abnormalities on CT or MRI brain imaging that may have an impact on the protocol compliance and/or PET scan
4. Patient who has dementia with MoCA-K ≤ 22
5. Patient who has a history of severe heart failure (NYHA class III to IV), stroke, cerebral ischemic attack, or seizure within 1 year prior to screening; or a history myocardial infarction or unstable angina within 6 months prior to screening.
6. Patient who has severe liver disease or has AST or ALT level 3 times more than ULN at the screening
7. Patient who has clinically significant depression [> 18 of Korean Beck Depression Inventory II score (K-BDI-II)]
8. Patient who has a history of brain surgery for any treatment of Parkinson's disease
9. Patient who has participated in any clinical trials for the treatment of Parkinson's Disease within 3 months prior to screening
10. Patient who took exenatide within 90 days prior to randomization
11. Patient who has a history of gastroduodenal ulcer or gastroparesis within 3 months prior to administration of investigational product or is currently on medication for acute or chronic gastritis
12. Patient who has severe kidney function injury (creatinine clearance < 30 ml/min)
13. Patient who has a history of pancreatitis
14. Patient who has type 1 or type 2 diabetes or HbA1c ≥ 6.5% at screening
15. Patient who has a history or suspected to thyroid cancer or multiple endocrine adenomatosis
16. Patient who has known or suspected intolerance in PET scan or fluoropropyl-CIT (18F)
17. Woman childbearing potential who doesn't agree to use the medically acceptable methods of contraception* during this study and up to 24 weeks after the last injection of investigational product

    *Medically acceptable methods of contraception: oral contraceptives, intrauterine contraceptive devices, vasectomy for male partner, barrier method [condom, spermicidal foam/gel/film/cream/suppository with sealed cap (diaphragm or cervix/bolt cap)].
18. Woman who is pregnant or breastfeeding
19. Patient who has a history of hypersensitivity reactions to any ingredients of investigational product
20. Patient who is not eligible for the study at the discretion of the investigator

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 99 (Estimated)
Dates: Start 2020-03-19 (Actual); Primary Completion 2021-09-29 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Change of MDS-UPDRS part 3 score | 48 week
  Change of MDS-UPDRS (Movement Disorder Society -Unified Parkinson's Disease Rating Scale ) part 3 score from baseline at 48 weeks.
  The MDS-UPDRS has four parts: Part I (non-motor experiences of daily living), Part II (motor experiences of daily living), Part III (motor examination) and Part IV (motor complications). The MDS-UPDRS consists of five measures, 0(normal) to 4(severe), according to each item, and is evaluated as the total score per part of Part 1 to 4. A 0 means there is no disability, and the higher the score, the more the disability is reflected.

SECONDARY OUTCOMES:
SNBR (specific to non-specific binding ratio) confirmed by PET scan | 0 and 48 weeks
  Change of SNBR (specific to non-specific binding ratio) from baseline at 48 weeks, confirmed by PET scan
MDS-UPDRS part 3 score | 0, 24 and 60 weeks
  Change of MDS-UPDRS (Movement Disorder Society -Unified Parkinson's Disease Rating Scale ) part 3 scores from baseline at 24 and 60 weeks.
  The MDS-UPDRS has four parts: Part I (non-motor experiences of daily living), Part II (motor experiences of daily living), Part III (motor examination) and Part IV (motor complications). The MDS-UPDRS consists of five measures, 0(normal) to 4(severe), according to each item, and is evaluated as the total score per part of Part 1 to 4. A 0 means there is no disability, and the higher the score, the more the disability is reflected.
MDS-UPDRS part 1, 2 and 4 scores | 0, 24, 48 and 60 weeks
  Changes of MDS-UPDRS (Movement Disorder Society -Unified Parkinson's Disease Rating Scale ) part 1, 2 and 4 scores from baseline at 24, 48 and 60 weeks.
  The MDS-UPDRS has four parts: Part I (non-motor experiences of daily living), Part II (motor experiences of daily living), Part III (motor examination) and Part IV (motor complications). The MDS-UPDRS consists of five measures, 0(normal) to 4(severe), according to each item, and is evaluated as the total score per part of Part 1 to 4. A 0 means there is no disability, and the higher the score, the more the disability is reflected.
K-PDQ-39 score | 0, 48 and 60 weeks
  Change of K-PDQ-39 (korean-The Parkinson's Disease Questionnaires-39) score from baseline at 48 and 60 weeks. PDQ-39 is an assessment of Parkinson's disease and comprises a total of 39 questions. Based on the past month's experience, each item consists of a five-point scale of 0(never) to 4 (always) and is checked by the test subjects themselves. The total score of PDQ-39 is evaluated as a percentage of 0-100%, and as the score increases, the symptom becomes more severe.
MoCA-K score | 0, 24, 48 and 60 weeks
  Change of MoCA-K (Montreal Cognitive Assessment-Korean) score from baseline at 24, 48 and 60 weeks.
  MoCA-K is designed to evaluate mild cognitive disorders. The raters evaluate cognitive functions such as attention and concentration, memory, language, conceptual thinking, calculations, and orientation. The execution time takes about 10 minutes and is evaluated by the sum of the scores of each item. A perfect score of 30 points or more is considered normal.
K-NMSS score | 0, 24, 48 and 60 weeks
  Change of K-NMSS (Korean-Non Motor Symptoms Scale) score from baseline at 24, 48 and 60 weeks.
  K-NMSS evaluates non-motorative symptoms of Parkinson's disease. It consists of a total of 30 questions, separated by nine aspects: cardiovascular function, sleep/ fatigue, sexual function, and other non-motor symptoms. The evaluation period is evaluated based on the experience of the last month.
  For each aspect, the grade point is evaluated as the degree of severity (level 0-3) and frequency (1-4), and the evaluation score is obtained by multiplying the degree and frequency of severity.
  The K-NMSS has a range of 0-360 points, and the higher the score, the more severe the symptoms are judged.
Each percentage of subjects and changing patterns in modified Hoehn and Yahr stage | 0, 24, 48 and 60 weeks
  Percentage of subjects per modified Hoehn and Yahr stage and the changing patterns from baseline at 24, 48 and 60 weeks
Change of the L-dopa dosage of subjects | 0, 2, 4, 8, 12, 24, 36, 48 and 60 weeks
  Starting time of L-dopa treatment and percentage of subjects who have L-dopa treatment at each visit.

OTHER OUTCOMES:
Pharmacokinetics test with blood | 0, 12, 24, 36, 48 and 60 weeks
  Pharmacokinetics test will assess Cmax (Maxi mum Plasma Concentration) and Tmax (Time of Maximum Plasma Concentration) in blood (pre-dose, 12, 24, 36, 48 and 60 weeks)
Pharmacokinetics test with CSF | 0, 12, 24, 36, 48 and 60 weeks
  Pharmacokinetics test will assess Cmax (Maximum Plasma Concentration) and Tmax (Time of Maximum Plasma Concentration) in Cerebrospinal Fluid (CSF; pre-dose and 48 weeks only)
Anti-exenatide antibodies test in blood | 0, 12, 24, 36, 48 and 60 weeks
  Check if antibody of exenatide (PT320) is created

CONTACTS AND LOCATIONS:
Overall Officials: Min Ho Ihm, Study Director — Peptron, Inc.
Locations (5):
- South Korea (5):
  - Seoul National University Bundang Hospital, Seongnam-si
  - Asan Medical Center, Seoul
  - Samsung Medical Center, Seoul
  - Seoul Metropolitan Government Seoul National University Boramae Medical Center, Seoul
  - Seoul National University Hospital, Seoul

IPD SHARING:
Plan to Share IPD: No